CLINICAL TRIAL: NCT00679991
Title: A Phase 1-2, Multi-Center, Dose Escalation Study of a Single Dose of PRT-201 Administered Immediately After Arteriovenous Fistula Creation in Patients With Chronic Kidney Disease
Brief Title: A Phase 1-2 Study of PRT-201 Administered in Chronic Kidney Disease (CKD) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Proteon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRT-201-101
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease
Keywords: arteriovenous fistula; AVF; hemodialysis; vascular access; PRT 201; dose escalation; dialysis; fistula; access; vonapanitase; kidney; renal
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula; Fistula | interventions — cholesterol-binding protein

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRT-201 (Active Comparator)
  Interventions: Drug: PRT-201
- 2 (Placebo Comparator)
  Interventions: Drug: PRT-201

INTERVENTIONS:
Drug: PRT-201 — Applied topically to AVF during surgery
  Arms: PRT-201
Drug: PRT-201 — Dose escalation study. Drug/placebo administered at the time of fistula creation

SUMMARY:
PRT-201 is a protein that causes long lasting dilation of blood vessels when applied to the outside surface of the blood vessel. The purpose of this study is to determine if PRT-201, when applied to a limited segment of blood vessel immediately after surgery to create an arteriovenous fistula (AVF), is safe, dilates the blood vessel, and increases blood flow through the AVF.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years.
* Chronic kidney disease with anticipated start of hemodialysis within six months or current hemodialysis dependence.
* Planned creation of a new AVF.

Exclusion Criteria:

* Patients for whom this is the only potential site for an AVF.
* By physical examination, absence of radial or ulnar artery flow or non-patent palmer arch.
* Treatment with any investigational agent within the previous 30 days or investigational antibody therapy within 90 days of signing informed consent.
* Pregnancy, lactation or plans to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a single topical dose of PRT-201. To assess the effect on the diameter of and blood flow through the AVF outflow vein. | 2 & 6 weeks after AVF creation

SECONDARY OUTCOMES:
The proportion of patients with AVF patency, AVF maturation, and AVF use for hemodialysis. | 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Clarian Health Partners/Indiana University/Purdue University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Western New England Renal & Transplant Associates, Springfield, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Methodist Hospital, Houston, Texas
  - Sentara Medical Group, Norfolk, Virginia

REFERENCES:
- [Result] Peden EK, Leeser DB, Dixon BS, El-Khatib MT, Roy-Chaudhury P, Lawson JH, Menard MT, Dember LM, Glickman MH, Gustafson PN, Blair AT, Magill M, Franano FN, Burke SK. A multi-center, dose-escalation study of human type I pancreatic elastase (PRT-201) administered after arteriovenous fistula creation. J Vasc Access. 2013 Apr-Jun;14(2):143-51. doi: 10.5301/jva.5000125. Epub 2012 Nov 20. PMID 23172172